CLINICAL TRIAL: NCT00042029
Title: A Double-Blind, Multicenter, Placebo-Controlled Study of MK0869 in the Treatment of Patients With Major Depressive Disorder
Brief Title: Treatment of Patients With Major Depressive Disorder With MK0869 (0869-073)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 0869-073; Formally-8DL718; MK0869-073; 2006_409
Record Dates: First submitted 2002-07-22; First posted 2002-07-23 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aprepitant

INTERVENTIONS:
Drug: MK0869, aprepitant
Drug: Comparator: placebo

SUMMARY:
A clinical study to determine the efficacy and safety of MK0869 in the treatment of depression.

DETAILED DESCRIPTION:
The duration of treatment is 8 weeks.

ELIGIBILITY:
Patients with Major Depressive Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2002-06-18 (Actual); Primary Completion 2003-10-03 (Actual); Study Completion 2003-10-03 (Actual)

PRIMARY OUTCOMES:
HAMD-17 total score; Tolerability

SECONDARY OUTCOMES:
CGI-I Scale score; Sheehan Disability Scale

REFERENCES:
- [Background] Keller M, Montgomery S, Ball W, Morrison M, Snavely D, Liu G, Hargreaves R, Hietala J, Lines C, Beebe K, Reines S. Lack of efficacy of the substance p (neurokinin1 receptor) antagonist aprepitant in the treatment of major depressive disorder. Biol Psychiatry. 2006 Feb 1;59(3):216-23. doi: 10.1016/j.biopsych.2005.07.013. Epub 2005 Oct 24. PMID 16248986
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html